CLINICAL TRIAL: NCT02834598
Title: Objectivating the Therapeutic Effect of a Rocking Movement by High Density Electroencephalography
Brief Title: Towards an Objectivation of the Therapeutic Effect of a Rocking Movement
Acronym: BAL-EASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: API/2012/27
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2016-07

CONDITIONS: Rocking Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rocking movement (Experimental): Participant is lying in a hammock with a rocking motion. Cerebral measurements from high-density electroencephalography while standard and deviant sounds are presented to the participant.
  Interventions: Device: high-density electroencephalography
- Lying position (Active Comparator): Participant is lying in a hammock with no rocking motion. Cerebral measurements from high-density electroencephalography while standard and deviant sounds are presented to the participant.
  Interventions: Device: high-density electroencephalography
- Seated position (Active Comparator): Participant is sitting on a chair. Cerebral measurements from high-density electroencephalography while standard and deviant sounds are presented to the participant.
  Interventions: Device: high-density electroencephalography

INTERVENTIONS:
Device: high-density electroencephalography — Cerebral measurements from high-density electroencephalography while standard and deviant sounds are presented to the participant.

SUMMARY:
The study evaluates the benefits of a rocking movement on well-being and attention, through high-density electroencephalography recordings. The effect of the rocking movement is compared to a seated position and a lying position.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* Informed consent

Exclusion Criteria:

* Pregnancy
* subjects with analgesic treatment
* subjects dependent on psychotropic substances

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Difference of amplitude between standard and deviant sounds | 20 minutes
  The amplitude of the mismatch negativity (corresponding to the difference between standard and deviant sounds) will be measured by electroencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: Régis Aubry, MD, PhD, Principal Investigator — Service douleur - soins palliatifs